CLINICAL TRIAL: NCT03171675
Title: Gingival Crevicular Fluid and Placental Tissue Levels of Interleukin-17 as a Possible Marker for Preterm Labor in Patients With Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Agoor, Principal Investigator, Ain Shams University
Other Study IDs: 22/01/2014; #33
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Chronic Periodontitis; Preterm Labor
Keywords: Chronic Periodontitis; Preterm Labor; Preterm Birth; Interleukin-17; IL-17; Periodontal Disease; Periodontitis; Periodontal risk factors; Medical risk factors
MeSH Terms: conditions — Chronic Periodontitis; Obstetric Labor, Premature; Premature Birth; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gingival crevicular fluid and placental tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Preterm/Chronic Periodontitis: Included ten female patients who underwent spontaneous preterm birth and were diagnosed with chronic periodontitis upon clinical examination
- Preterm/Healthy Periodontium: Included ten female patients who underwent spontaneous preterm birth and who had a healthy periodontium upon clinical examination
- Term/Chronic Periodontitis: Included ten female patients who underwent spontaneous normal term birth and were diagnosed with chronic periodontitis upon clinical examination
- Term/Healthy Periodontium: Included ten female patients who underwent spontaneous normal term birth and who had a healthy periodontium upon clinical examination (Armitage1999)

SUMMARY:
This case control-study measures the levels of Interleukin-17 in gingival crevicular fluid and placental tissue samples of pregnant females as a possible marker in determining whether or not an association exists between chronic periodontitis and preterm labor. Interleukin-17 is a pro-inflammatory cytokine whose levels have been proven to increase in periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

1. Within the age range of 18-35 years
2. Free of any systemic diseases as referenced from Burket's Oral Medicine health history questionnaire (Glick2008)
3. Spontaneous normal term birth at ≥37 weeks of gestation without any obstetrical or medical complications
4. Spontaneous preterm birth (PTB) at <37 weeks of gestation after uterine contraction or rupture of membranes (Keelan1999)

Exclusion Criteria:

1. History of medications that may affect the study outcome, such as: current use of systemic corticosteroids or antibiotics for at least one month
2. Genital and urinary tract infections
3. Existing hypertension and diabetes mellitus before pregnancy, autoimmune disease, asthma, and chronic renal disease
4. Multiple pregnancies, cervical cerculage, abnormal placentation, past history of preterm delivery, or antepartum hemorrhage
5. Low or high maternal body mass index

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Conducted in Cairo, Egypt at the Maternal-Fetal Medical Clinic at the Department of Obstetrics and Gynecology, Faculty of Medicine, Ain Shams University.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-12-25 (Actual); Primary Completion 2015-03-02 (Actual); Study Completion 2015-06-16 (Actual)

PRIMARY OUTCOMES:
Interleukin-17 | Single sample from each patient following birth
  Interleukin-17 levels in gingival crevicular fluid and placental tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y. Gamal, PhD, Study Chair — Faculty of Dentistry, Ain Shams University; Olfat G. Shaker, PhD, Study Director — Cairo University; Fatma H. Mohamed, PhD, Study Director — Faculty of Dentistry, Ain Shams University; Mohamed Agoor, MSc, Principal Investigator — Faculty of Dentistry, Ain Shams University

REFERENCES:
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Glick M, Greenberg MS, Ship JA. Introduction to oral medicine and oral diagnosis: evaluation of the dental patient. In: Greenberg MS, Glick M, Ship JA. Burket's Oral Medicine. 11th Edition. Hamilton, Ontario: BC Decker; 2008:3.
- [Background] Keelan JA, Marvin KW, Sato TA, Coleman M, McCowan LM, Mitchell MD. Cytokine abundance in placental tissues: evidence of inflammatory activation in gestational membranes with term and preterm parturition. Am J Obstet Gynecol. 1999 Dec;181(6):1530-6. doi: 10.1016/s0002-9378(99)70400-x. PMID 10601939